CLINICAL TRIAL: NCT04197284
Title: Comparison of Efficacy of Biofeedback, Electrical Stimulation and Therapeutic Exercise in Patients With Knee Osteoarthritis
Brief Title: Determination of the Effectiveness of Certain Physical Methods in the Treatment of Knee Osteoarthritis
Acronym: BFBOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Silvija Mahnik, MD, Physical medicine and rehabilitation specialist, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1505984
Record Dates: First submitted 2019-11-10; First posted 2019-12-13 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; biofeedback; electrical stimulation; kinesitherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Biofeedback, Psychology; Electric Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research will be single-blind. Randomization of patients will be performed immediately prior to physical therapy using web page www.randomization.com, and the results of the randomization will be known to the physician who will not be directly involved in the treatment or examination of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): In control group subjects will undergo individual kinesitherapy- isometric exercise for strengthening of the quadriceps muscle.
  Interventions: Other: kinesitherapy
- Biofeedback group (Active Comparator): Biofeedback group will perform physical therapy using biofeedback device for better activation control of the quadriceps muscle with audio and visual signal. They will also perform isometric exercise.
  Interventions: Device: Biofeedback, Myomed 632; Other: kinesitherapy
- Electrical stimulation (Active Comparator): Electrical stimulation group will receive electrical stimulation of the quadriceps muscle and they will also perform isometric exercise.
  Interventions: Device: device for electrical stimulation, BTL 4000 Smart; Other: kinesitherapy

INTERVENTIONS:
Device: Biofeedback, Myomed 632 — Biofeedback is a mind-body technique that involves using visual or auditory feedback to gain control over involuntary bodily functions.
  Electrical stimulation is a technique used to elicit a muscle contraction using electrical impulses.
  Arms: Biofeedback group
Device: device for electrical stimulation, BTL 4000 Smart — Electrical stimulation is a technique used to elicit a muscle contraction using electrical impulses. Electrodes, controlled by a unit, are placed on the skin over a predetermined area. Electrical current is then sent from the unit to the electrodes and delivered into the muscle causing a contraction.
  Arms: Electrical stimulation
Other: kinesitherapy — isometric exercise of the quadriceps muscle

SUMMARY:
Osteoarthritis (OA) is a chronic joint disease that involves the entire joint, causing cartilage damage, bone remodeling, osteophyte formation and loss of normal joint function. Knee OA is one of the leading causes of disability in the world and thus represents a major public health problem. Knee OA treatment can be operative and non-operative. Non-operative treatment includes pharmacological treatment, changing life style and physical therapy. The goal of physical therapy in knee OA is to reduce pain and improve knee function through therapeutic exercise, especially by strengthening the quadriceps muscle. In addition to therapeutic exercise, muscle electrical stimulation is often used, and in the literature there is evidence of biofeedback therapy efficacy.

Goal of the study is to investigate whether there is a difference in pain reduction, increase in quadriceps muscle strength, and improvement in knee function in patients who had only kinesitherapy, from those who underwent kinesitherapy and biofeedback, and in patients who received electrical stimulation of quadriceps muscle with kinesitherapy. 93 patients with knee OA according to ACR criteria and Kellgren and Lawrence radiological classification grades 1 and 2 will be included in study. Subjects will complete: Visually Analogous Pain Scale (VAS), Western Ontario Universities Osteoarthritis Index (WOMAC), 36 Item Short Form Health Survey (SF 36), International Classification of Functioning, Disability and Health (ICF) osteoarthritis core set, and quadriceps muscle strength will be measured by EMG biofeedback device.

DETAILED DESCRIPTION:
The research will be conducted in the Department of Orthopedic surgery of the Clinical Hospital Center Zagreb. The research will be prospective, randomized, single blinded. Randomization of patients will be performed before physical therapy using web site www.randomization.com, and the results of the randomization will be known to the physician who will not be directly involved in the treatment or examination of patients.

All patients will sign informed consent before the study begins. Research has been approved by the Ethics Committee of Clinical Hospital Center Zagreb and Ethics committee of the School of Medicine, University of Zagreb.

Inclusion criteria are: patients age 55 years and older who have knee OA according to the American College of Rheumatology criteria (ACR) and knee OA according to Kellgren and Lawrence Radiology Classification Grade 1 and 2, and who report knee pain for at least 3 months. Exclusion criteria are: patients who had surgery on that knee, patients with a pacemaker, and metallic foreign body in the area of muscle stimulation, patients with thrombophlebitis and deep vein thrombosis, patients with skin infection, malignancy, bleeding disorders, patients with neurological disease, patients with inflammatory rheumatological disease, with congenital and acquired knee deformities, with contractures of the hips and ankles, with grade 3 and 4 osteoarthritis according to Kellgren and Lawrence classification, patients who received intraarticular knee injection in the last 3 months and patients with post-traumatic knee osteoarthritis and osteonecrosis.

The investigators will record: age, sex, height, weight, body mass index, leg length and use of orthopedics aids. Clinical examination will be performed on the first day, day 21, after 90 and after 180 days.

At each examination patients will complete following questionnaires: Visually Analog Scale for pain (VAS), Western Ontario Universities Osteoarthritis Index (WOMAC), 36 Item Short Form Health Survey (SF 36) and International Classification of Functioning, Disability and Health (ICF) osteoarthritis core set.

Quadriceps muscle strength will be measured with a Biofeedback therapy device (EMG Biofeedback, Myomed 632, United Kingdom, 2017) .

Patients will be randomisen in three groups. Patients in the first group will be treated with individual kinesitherapy. Patients in the second group will be treated with individual kinesitherapy and biofeedback therapy for strengthening of the quadriceps muscle using EMG Biofeedback device, Myomed 632, United Kingdom, 2017.

Patients in the third group will be treated with individual kinesitherapy together with electrical stimulation of the quadriceps muscle using electrostimulation device (BTL- 4000 Smart, United Kingdom, 2017).

The required sample size was calculated based on pain values data reported in the study by Choi et al. Pain was measured using VAS scale, and sample size was calculated using G Power software package (v3.1.9.4). With the parameter of statistical significance level (alpha) of 0.05 and a test power (1 - beta) of 0.90, based on the data from the Choi et al work, the required final sample size is a total of 93 subjects and 31 subjects for each of the three groups.

The investigators expect to find that kinesitherapy and biofeedback therapy are more efficient compared to kinesitherapy alone or and kinesitherapy and electrical stimulation in reducing pain, improving knee function and strengthening of the quadriceps muscle.

ELIGIBILITY:
Inclusion Criteria:

* radiological evidence of primary OA with Grade 1 and 2 on the Kellgren-Lawrence Scale
* knee pain for 3 months
* knee osteoarthritis defined by American College of Rheumatology Criteria

Exclusion Criteria:

* surgery on that knee
* pacemaker
* metallic foreign body in the area of stimulation
* thrombophlebitis and thrombosis
* skin infection
* malignancy,
* bleeding disorders
* neurological disease
* inflammatory rheumatology disease
* congenital and acquired knee deformities
* contracture of the hips and ankles
* grade 3 and 4 osteoarthritis om the Kellgren and Lawrence classification
* intraarticular injection in the last 3 months
* post-traumatic knee osteoarthritis and osteonecrosis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Impact of biofeedback therapy on change in knee pain measured on Visual Analogue Scale (VAS). | 3 weeks
  Determine whether the use of biofeedback for quadriceps muscle strengthening will change knee pain score measured on Visual Analogue Scale (VAS). Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of biofeedback therapy on change in knee pain measured on Visual Analogue Scale (VAS). | 3 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening will change knee pain score measured on Visual Analogue Scale (VAS). Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of biofeedback therapy on change in knee pain measured on Visual Analogue Scale (VAS). | 6 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening will change knee pain score measured on Visual Analogue Scale (VAS). Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Impact of biofeedback therapy on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 weeks
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of biofeedback therapy on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of biofeedback therapy on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 6 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of biofeedback therapy on muscle strength measured by EMG biofeedback device. | 3 weeks
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of biofeedback therapy on muscle strength measured by EMG biofeedback device. | 3 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of biofeedback therapy on muscle strength measured by EMG biofeedback device. | 6 months
  Determine whether the use of biofeedback for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of kinesitherapy on knee pain measured on Visual Analogue Scale (VAS). | 3 weeks
  Determine whether kinesitherapy for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of kinesitherapy on knee pain measured on Visual Analogue Scale (VAS). | 3 months
  Determine whether kinesitherapy for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of kinesitherapy on knee pain measured on Visual Analogue Scale (VAS). | 6 months
  Determine whether kinesitherapy for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of kinesitherpay on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 weeks
  Determine whether kinesitherapy for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of kinesitherpay on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 months
  Determine whether kinesitherapy for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of kinesitherpay on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 6 months
  Determine whether kinesitherapy for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of kinesiotherapy on quadriceps muscle strength measured by EMG biofeedback device. | 3 weeks
  Determine whether kinesitherapy for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of kinesiotherapy on quadriceps muscle strength measured by EMG biofeedback device. | 3 months
  Determine whether kinesitherapy for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of kinesiotherapy on quadriceps muscle strength measured by EMG biofeedback device. | 6 months
  Determine whether kinesitherapy for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of electrical stimulation of the quadriceps muscle on knee pain measured on Visual Analogue Scale (VAS). | 3 weeks
  Determine whether electrical stimulation for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of electrical stimulation of the quadriceps muscle on knee pain measured on Visual Analogue Scale (VAS). | 3 months
  Determine whether electrical stimulation for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of electrical stimulation of the quadriceps muscle on knee pain measured on Visual Analogue Scale (VAS). | 6 months
  Determine whether electrical stimulation for quadriceps muscle strengthening will change knee pain score measured on VAS scale. Change will be measured on VAS scale in millimeters, from 0 to 100 mm, a higher score indicates greater pain intensity.
Impact of electrical stimulation on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 weeks
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of electrical stimulation on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 3 months
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of electrical stimulation on knee function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC). | 6 months
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes knee function score measured by WOMAC questionnaire. Questionnaire consists 24 items divided into 3 subscales: Pain, Stifness and Physical Functioning. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.The test questions are scored on a scale of 0-4 , from best to worse. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Impact of electrical stimulation on quadriceps muscle strength measured by EMG biofeedback device. | 3 weeks
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of electrical stimulation on quadriceps muscle strength measured by EMG biofeedback device. | 3 months
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.
Impact of electrical stimulation on quadriceps muscle strength measured by EMG biofeedback device. | 6 months
  Determine whether the use of electrical stimulation for quadriceps muscle strengthening changes quadriceps muscle strength measured on EMG biofeedback device in micro volts during maximal voluntary isometric contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bojanić, Prof Phd, Study Chair — Universty of Zagreb, School of medicine
Locations (1):
- University Hospital Centre Zagreb, Department of Orthopaedic Surgery, Zagreb, Croatia

REFERENCES:
- [Background] Choi YL, Kim BK, Hwang YP, Moon OK, Choi WS. Effects of isometric exercise using biofeedback on maximum voluntary isometric contraction, pain, and muscle thickness in patients with knee osteoarthritis. J Phys Ther Sci. 2015 Jan;27(1):149-53. doi: 10.1589/jpts.27.149. Epub 2015 Jan 9. PMID 25642061
- [Background] Lucca JA, Recchiuti SJ. Effect of electromyographic biofeedback on an isometric strengthening program. Phys Ther. 1983 Feb;63(2):200-3. doi: 10.1093/ptj/63.2.200. PMID 6823470
- [Background] Yilmaz OO, Senocak O, Sahin E, Baydar M, Gulbahar S, Bircan C, Alper S. Efficacy of EMG-biofeedback in knee osteoarthritis. Rheumatol Int. 2010 May;30(7):887-92. doi: 10.1007/s00296-009-1070-9. Epub 2009 Aug 20. PMID 19693508
- [Background] Akkaya N, Ardic F, Ozgen M, Akkaya S, Sahin F, Kilic A. Efficacy of electromyographic biofeedback and electrical stimulation following arthroscopic partial meniscectomy: a randomized controlled trial. Clin Rehabil. 2012 Mar;26(3):224-36. doi: 10.1177/0269215511419382. Epub 2011 Oct 4. PMID 21971752
- [Background] Raeissadat SA, Rayegani SM, Sedighipour L, Bossaghzade Z, Abdollahzadeh MH, Nikray R, Mollayi F. The efficacy of electromyographic biofeedback on pain, function, and maximal thickness of vastus medialis oblique muscle in patients with knee osteoarthritis: a randomized clinical trial. J Pain Res. 2018 Nov 8;11:2781-2789. doi: 10.2147/JPR.S169613. eCollection 2018. PMID 30519081
- [Background] Cherian JJ, McElroy MJ, Kapadia BH, Bhave A, Mont MA. Prospective Case Series of NMES for Quadriceps Weakness and Decrease Function in Patients with Osteoarthritis of the Knee. J Long Term Eff Med Implants. 2015;25(4):301-6. doi: 10.1615/jlongtermeffmedimplants.2015012620. PMID 26852638
- [Background] Giggins O, Fullen B, Coughlan G. Neuromuscular electrical stimulation in the treatment of knee osteoarthritis: a systematic review and meta-analysis. Clin Rehabil. 2012 Oct;26(10):867-81. doi: 10.1177/0269215511431902. Epub 2012 Feb 9. PMID 22324059
- [Background] Durmus D, Alayli G, Canturk F. Effects of quadriceps electrical stimulation program on clinical parameters in the patients with knee osteoarthritis. Clin Rheumatol. 2007 May;26(5):674-8. doi: 10.1007/s10067-006-0358-3. Epub 2006 Aug 1. PMID 16897119
- [Background] de Oliveira Melo M, Aragao FA, Vaz MA. Neuromuscular electrical stimulation for muscle strengthening in elderly with knee osteoarthritis - a systematic review. Complement Ther Clin Pract. 2013 Feb;19(1):27-31. doi: 10.1016/j.ctcp.2012.09.002. Epub 2012 Oct 18. PMID 23337561
- [Background] de Oliveira Melo M, Pompeo KD, Baroni BM, Vaz MA. Effects of neuromuscular electrical stimulation and low-level laser therapy on neuromuscular parameters and health status in elderly women with knee osteoarthritis: A randomized trial. J Rehabil Med. 2016 Mar;48(3):293-9. doi: 10.2340/16501977-2062. PMID 26871692
- [Background] Zeng C, Li H, Yang T, Deng ZH, Yang Y, Zhang Y, Lei GH. Electrical stimulation for pain relief in knee osteoarthritis: systematic review and network meta-analysis. Osteoarthritis Cartilage. 2015 Feb;23(2):189-202. doi: 10.1016/j.joca.2014.11.014. Epub 2014 Nov 26. PMID 25497083
- [Background] Lepley AS, Gribble PA, Pietrosimone BG. Effects of electromyographic biofeedback on quadriceps strength: a systematic review. J Strength Cond Res. 2012 Mar;26(3):873-82. doi: 10.1519/JSC.0b013e318225ff75. PMID 22289696
- [Background] Eid MA, Aly SM, El-Shamy SM. Effect of Electromyographic Biofeedback Training on Pain, Quadriceps Muscle Strength, and Functional Ability in Juvenile Rheumatoid Arthritis. Am J Phys Med Rehabil. 2016 Dec;95(12):921-930. doi: 10.1097/PHM.0000000000000524. PMID 27149595
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Grazio S. [International Classification of Functioning, Disability and Health (ICF) in the most important diseases and conditions of rheumatology practice]. Reumatizam. 2011;58(1):27-43. Croatian. PMID 21751573
- [Background] Maslic Sersic D, Vuletic G. Psychometric evaluation and establishing norms of Croatian SF-36 health survey: framework for subjective health research. Croat Med J. 2006 Feb;47(1):95-102. PMID 16489702
- [Background] Hurley MV, Scott DL. Improvements in quadriceps sensorimotor function and disability of patients with knee osteoarthritis following a clinically practicable exercise regime. Br J Rheumatol. 1998 Nov;37(11):1181-7. doi: 10.1093/rheumatology/37.11.1181. PMID 9851266